CLINICAL TRIAL: NCT00705536
Title: A Phase I, Randomized, Double-Blind Crossover Pharmacokinetic, Pharmacodynamic, and Safety Study of Subcutaneously Administered Humalog® (Insulin Lispro Injection; Rapid-Acting Insulin) With and Without Recombinant Human Hyaluronidase (rHuPH20) Versus Subcutaneously Administered Humulin R® (Regular Insulin Injection) With and Without rHuPH20
Brief Title: Pharmacokinetic (PK), Pharmacodynamic (PD), and Safety Study of Subcutaneously Administered Humalog® With and Without Recombinant Human Hyaluronidase (rHuPH20)and Humulin-R® With and Without rHuPH20
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HZ2-07-04
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: rHuPH20; Hyaluronidase; Insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro; Insulin; Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Humalog first, then Humalog + rHuPH20 (Active Comparator): Humalog first, then Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
  A single subcutaneous (SC) injection of 20 units (U) Humalog on Day 1 of the study, followed by a single SC injection of 20 U Humalog + 300 U rHuPH20 after a washout period of at least 6 days
  Interventions: Drug: Humalog; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humalog + rHuPH20 first, then Humalog (Active Comparator): Humalog + recombinant human hyaluronidase PH20 (rHuPH20) first, then Humalog
  A single subcutaneous (SC) injection of 20 units (U) Humalog + 300 U rHuPH20 on Day 1 of the study, followed by a single SC injection of 20 U Humalog after a washout period of at least 6 days
  Interventions: Drug: Humalog; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humulin-R first, then Humulin-R + rHuPH20 (Active Comparator): Humulin-R (recombinant human insulin) first, then Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
  A single subcutaneous (SC) injection of 20 units (U) Humulin-R on Day 1 of the study, followed by a single SC injection of 20 U Humulin-R + 240 U rHuPH20 after a washout period of at least 6 days
  Interventions: Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humulin-R + rHuPH20 first, then Humulin-R (Active Comparator): Humulin-R (recombinant human insulin) + recombinant human hyaluronidase PH20 (rHuPH20) first, then Humulin-R
  A single subcutaneous (SC) injection of 20 units (U) Humulin-R + 240 U rHuPH20 on Day 1 of the study, followed by a single SC injection of 20 U Humulin-R after a washout period of at least 6 days
  Interventions: Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)

INTERVENTIONS:
Drug: Humalog
  Other Names: Insulin lispro
  Arms: Humalog + rHuPH20 first, then Humalog; Humalog first, then Humalog + rHuPH20
Drug: Humulin-R
  Other Names: Humulin; Recombinant human insulin
  Arms: Humulin-R + rHuPH20 first, then Humulin-R; Humulin-R first, then Humulin-R + rHuPH20
Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: PH20; HYLENEX

SUMMARY:
The purpose of the study is to compare the pharmacokinetics (PK) and pharmacodynamics (PD) of Humalog (insulin lispro) or Humulin-R (recombinant human insulin) when administered as a single subcutaneous (SC) injection of 20 units (U) with or without coadministration of recombinant human hyaluronidase PH20 (rHuPH20).

The study hypothesizes that the time required to reach maximum insulin concentration (tmax) when insulin is administered with rHuPH20 will be comparable or shorter than the time required without rHuPH20.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male participants aged 18 to 55 years.
2. Body mass index (BMI) 18 to 28 kilograms per meter squared (kg/m^2) and total body weight >70 kilograms (kg) (154 pounds [lb]).
3. Willingness and ability to comply with the protocol.
4. Vital signs within the normal range.
5. Within 7 days before the first injection, metabolic panel results and complete blood count (CBC) within the laboratory normal reference range.
6. Fasting plasma glucose within the normal range of 90 to 110 milligrams per deciliter (mg/dL) on the morning of the glucose clamp.
7. Agreement not to father a child or donate sperm and to use effective contraception during the study and for at least 30 days after study completion.
8. Willingness and ability to sign an informed consent form.

Exclusion Criteria:

1. Evidence or history of clinically significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic (to include history of seizures) or allergic disease, or history of hypoglycemic episodes.
2. Known history of diabetes mellitus.
3. Prior exposure to any insulin or insulin analogs.
4. Known allergy to hyaluronidase or any other ingredient in HYLENEX.
5. Known allergy to bee or vespid venom.
6. Positive urine drug screen results.
7. Positive human immunodeficiency virus (HIV) 1, HIV 2, hepatitis B, or hepatitis C antibody test result.
8. Any history or evidence of alcohol or drug abuse.
9. History or evidence of use of any tobacco- or nicotine-containing product within 6 months of screening, or screening urine nicotine concentration >50 nanograms per milliliter (ng/mL).
10. Use of prescription or nonprescription drugs within 7 days or 5 half-lives, whichever was shorter, except acetaminophen at doses of less than or equal to 1 gram per day (g/day).
11. Donation of blood in excess of 500 milliliters (mL) within 56 days before dosing.
12. Failure to limit alcohol consumption and refrain from exercise within 48 hours before each injection.
13. Known clinically significant intercurrent illness or other major systemic disease that would unduly risk the participant's safety or interfere with the interpretation of results.
14. Participation in a study of any investigational drug or device 30 days before enrollment in this study.
15. Unfitness for the study, in the investigator's opinion.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Kipnes, MD, Principal Investigator — Diabetes and Glandular Disease Research Associates Inc.
Locations (1):
- Diabetes and Glandular Disease Research, Inc., San Antonio, Texas, United States

REFERENCES:
- [Result] Vaughn DE, Yocum RC, Muchmore DB, Sugarman BJ, Vick AM, Bilinsky IP, Frost GI. Accelerated pharmacokinetics and glucodynamics of prandial insulins injected with recombinant human hyaluronidase. Diabetes Technol Ther. 2009 Jun;11(6):345-52. doi: 10.1089/dia.2009.0013. PMID 19459762

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Humalog First, Then Humalog + rHuPH20: Stage 1 of the study: A single subcutaneous (SC) injection of 20 units (U) Humalog alone on Day 1 of Stage 1, followed by a washout period of at least 6 days. Then, a single SC injection of 20 U Humalog + 300 U recombinant human hyaluronidase PH20 (rHuPH20).
- Stage 1: Humalog + rHuPH20 First, Then Humalog: Stage 1 of the study: A single subcutaneous (SC) injection of 20 units (U) Humalog + 300 U recombinant human hyaluronidase PH20 (rHuPH20) on Day 1 of Stage 1, followed by a washout period of at least 6 days. Then, a single SC injection of 20 U Humalog alone.
- Stage 2: Humulin-R First, Then Humulin-R + rHuPH20: Stage 2 of the study: A single subcutaneous (SC) injection of 20 units (U) Humulin-R alone on Day 1 of Stage 2, followed by a washout period of at least 6 days. Then, a single SC injection of 20 U Humulin-R + 240 U recombinant human hyaluronidase PH20 (rHuPH20).
- Stage 2: Humulin-R + rHuPH20 First, Then Humulin-R: Stage 2 of the study. A single subcutaneous (SC) injection of 20 units (U) Humulin-R + 240 U recombinant human hyaluronidase PH20 (rHuPH20) on Day 1 of Stage 2, followed by a washout period of at least 6 days. Then, a single SC injection of 20 U Humulin-R alone.
Period: Start Period 1
Arm/Group | Stage 1: Humalog First, Then Humalog + rHuPH20 | Stage 1: Humalog + rHuPH20 First, Then Humalog | Stage 2: Humulin-R First, Then Humulin-R + rHuPH20 | Stage 2: Humulin-R + rHuPH20 First, Then Humulin-R
Started | 6 | 6 | 7 | 7
Received at Least 1 Dose of Study Drug | 6 | 6 | 7 | 7
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Washout Period of at Least 6 Days
Arm/Group | Stage 1: Humalog First, Then Humalog + rHuPH20 | Stage 1: Humalog + rHuPH20 First, Then Humalog | Stage 2: Humulin-R First, Then Humulin-R + rHuPH20 | Stage 2: Humulin-R + rHuPH20 First, Then Humulin-R
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Start Period 2
Arm/Group | Stage 1: Humalog First, Then Humalog + rHuPH20 | Stage 1: Humalog + rHuPH20 First, Then Humalog | Stage 2: Humulin-R First, Then Humulin-R + rHuPH20 | Stage 2: Humulin-R + rHuPH20 First, Then Humulin-R
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Completed Study
Arm/Group | Stage 1: Humalog First, Then Humalog + rHuPH20 | Stage 1: Humalog + rHuPH20 First, Then Humalog | Stage 2: Humulin-R First, Then Humulin-R + rHuPH20 | Stage 2: Humulin-R + rHuPH20 First, Then Humulin-R
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of Humalog or Humulin-R with or without rHuPH20.
Groups:
- Stage 1: Humalog Alone or Humalog + rHuPH20: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humalog alone or 20 U Humalog + 300 U recombinant human hyaluronidase (rHuPH20), followed by crossover treatment after a washout period of at least 6 days.
- Stage 2: Humulin-R Alone or Humulin-R + rHuPH20: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humulin-R alone or 20 U Humulin-R + 240 U recombinant human hyaluronidase (rHuPH20), followed by crossover treatment after a washout period of at least 6 days.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Humalog Alone or Humalog + rHuPH20 | Stage 2: Humulin-R Alone or Humulin-R + rHuPH20 | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (7.8) | 36.7 (8.9) | 37.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximum Serum Insulin Concentration (Tmax)
Description: Time to maximum serum insulin concentration (tmax) values for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from 3 milliliter (mL) blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable tmax data.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Stage 1: Humalog Alone: Humalog: A single subcutaneous (SC) injection of 20 units (U)
- Stage 1: Humalog + rHuPH20: Humalog + recombinant human hyaluronidase PH20 (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) Humalog and 300 U rHuPH20
- Stage 2: Humulin-R Alone: Humulin-R: A single subcutaneous (SC) injection of 20 units (U)
- Stage 2: Humulin-R + rHuPH20: Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) Humulin-R and 240 U rHuPH20
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Minutes | 97.5 (35.9) | 48.0 (7.99) | 163 (51.5) | 67.8 (19.1)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0006, ANOVA — Treatment comparison of Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0002, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

2. Primary Outcome: Maximum Serum Insulin Concentration (Cmax)
Description: Maximum serum insulin concentration (Cmax) values for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from 3 milliliter (mL) blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable Cmax data.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Picomoles per liter | 680 (361) | 1290 (471) | 390 (137) | 944 (257)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0003, ANOVA — Treatment comparison of Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

3. Secondary Outcome: Time to Maximum Glucose Infusion Rate (tGIR[Max])
Description: Time to maximal effect for glucose infusion rate (tGIR[max]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from blood samples obtained every 3 minutes during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable tGIR(max) data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Minutes | 193 (58.2) | 114 (43.0) | 253 (61.8) | 165 (51.2)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0059, ANOVA — Treatment comparison of Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0105, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

4. Secondary Outcome: Time to Early Half-Maximal Effect for Glucose Infusion Rate (tGIR[early50%])
Description: Time to early half-maximal effect for glucose infusion rate (tGIR[early50%]) for participants who were randomized to Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable tGIR(early50%) data.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Stage 1. Humalog Alone: Humalog: A single subcutaneous (SC) injection of 20 units (U)
- Stage 1: Humalog + rHuPH20: Humalog + recombinant human hyaluronidase PH20 (rHuPH20) : A single subcutaneous (SC) injection of 20 units (U) Humalog + 300 U rHuPH20
Arm/Group | Stage 1. Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Minutes | 72.3 (16.6) | 43.8 (15.1) | 104 (33.3) | 47.4 (13.1)
Statistical Analysis 1: Comparison: Stage 1. Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0002, ANOVA — Treatment comparison for Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

5. Secondary Outcome: Time to Late Half-Maximal Effect for Glucose Infusion Rate (tGIR[late50%])
Description: Time to late half-maximal effect for glucose infusion rate (tGIR[late50%]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) were measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
  Because the study was only 360 minutes in duration, there was not sufficient time for regular human insulin to show an effect and therefore tGIR(late50%) could not be calculated for participants receiving Humulin-R alone.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, or Humulin-R + rHuPH20 with evaluable tGIR(late50%) data.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Stage 1: Humalog + rHuPH20: Humalog + recombinant human hyaluronidase (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) Humalog and 300 U rHuPH20
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13
Minutes | 324 (32.9) | 275 (48.0) | 282 (68.0)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.3019, ANOVA — Treatment comparison for Humalog alone and Humalog + rHuPH20 using a pairwise t-test

6. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to the Time Required to Reach Endogenous Plasma Glucose Levels (AUC[0-t'])
Description: Area under the serum concentration-time curve from time zero to the time required to reach endogenous plasma glucose levels (AUC[0-t']) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from 3 milliliter (mL) blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(0-t') data.
Measure: Mean (Standard Deviation); unit: Picomoles per liter times minutes
Groups:
- Stage 2: Humulin-R + rHuPH20: Humulin + recombinant human hyaluronidase PH20 (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) Humulin-R and 240 U rHuPH20
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Picomoles per liter times minutes | 116000 (23000) | 133000 (21800) | 91400 (25700) | 137000 (32800)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0401, ANOVA — Treatment comparison of Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0004, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

7. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time to Reach Maximum Concentration (Tmax) for Serum Insulin With Recombinant Human Hyaluronidase PH20 (rHuPH20) (AUC[0-tmaxPH20])
Description: Area under the concentration-time curve from time 0 to time to reach maximum concentration (tmax) for serum insulin (Humalog or Humulin-R) with recombinant human hyaluronidase (rHuPH20) (AUC[0-tmaxPH20]) for participants who received Humalog or Humulin-R and with rHuPH20 were measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment and every 3 min from min 0 through 48 for Stage 1 and, and every 3 min from min 0 through 68 for Stage 2 during the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 48 minutes postdose during Stage 1, or up to 68 minutes postdose during Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(0-tmaxPH20) data.
Measure: Mean (Standard Deviation); unit: Picomoles per liter times minutes
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Picomoles per liter times minutes | 9530 (10500) | 27900 (14300) | 8780 (3010) | 34800 (9150)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — Treatment comparison of Humalog alone and Humalog +rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

8. Primary Outcome: Relative Bioavailability (Area Under the Curve [AUC] for Insulin + Recombinant Human Hyaluronidase [rHuPH20] / AUC for Insulin Alone)
Description: Relative bioavailability was determined by dividing the baseline-corrected geometric mean of the area under the curve (AUC) for insulin (ins) (Humalog or Humulin-R) with recombinant human hyaluronidase PH20 (rHuPH20) by the baseline-corrected geometric mean of the AUC for insulin alone (AUC[insulin+rHuPH20]/AUC[insulin]).
  Bioavailability values for participants who received Humalog or Humulin-R and rHuPH20 were measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog + rHuPH20 or Humulin-R + rHuPH20 with evaluable relative bioavailability (AUC[insulin+rHuPH20]/AUC[insulin alone]) data.
Measure: Mean (Standard Deviation); unit: Ratio of AUC(ins+rHuPH20)/AUC(ins alone)
Groups:
- Stage 1: Humalog + rHuPH20: Humalog + recombinant human hyaluronidase (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) of Humalog and 300 U of rHuPH20
- Stage 2: Humulin-R + rHuPH20: Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20): A single subcutaneous (SC) injection of 20 units (U) of Humulin-R and 240 U of rHuPH20
Arm/Group | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 13
Ratio of AUC(ins+rHuPH20)/AUC(ins alone) | 1.18 (0.221) | 1.57 (0.406)

9. Secondary Outcome: Maximum Glucose Infusion Rate (GIR[Max])
Description: Maximum glucose infusion rate (GIR[max]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase PH20 (rHuPH20) were measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 through 360 throughout the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable GIR(max) data.
Measure: Mean (Standard Deviation); unit: Milligrams per kilogram per minute
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Milligrams per kilogram per minute | 8.11 (4.48) | 8.57 (4.24) | 7.82 (2.52) | 10.5 (3.89)
Statistical Analysis 1: Comparison: Stage 1: Humalog Alone vs Stage 1: Humalog + rHuPH20; Test type: Superiority or Other; p = 0.5589, ANOVA — Treatment comparison of Humalog alone and Humalog + rHuPH20 using a pairwise t-test
Statistical Analysis 2: Comparison: Stage 2: Humulin-R Alone vs Stage 2: Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0067, ANOVA — Treatment comparison of Humulin-R alone and Humulin-R + rHuPH20 using a pairwise t-test

10. Secondary Outcome: Area Under the Glucose Infusion Rate Curve From 0 to 60 Minutes After Injection (AUC[GIR{0-60}])
Description: The area under the curve for the glucose infusion rate from minutes (min) 0 to 60 after injection (AUC[GIR{0-60}]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) was measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 min prior to treatment and every 3 min from min 0 through 60 during the clamp procedure. Means were calculated using analysis of variance with fixed of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 60 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(GIR[0-60]) data.
Measure: Mean (Standard Deviation); unit: Grams per kilogram
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Grams per kilogram | 82.8 (51.9) | 167 (81.0) | 74.3 (40.4) | 180 (57.7)

11. Secondary Outcome: Area Under the Glucose Infusion Rate Curve From 0 to 120 Minutes After Injection (AUC[GIR{0-120}])
Description: The area under the glucose infusion rate curve from minutes 0 to 120 after injection (AUC[GIR{0-120}]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) was measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 minute (min) prior to treatment, every 3 min from min 0 through 60, and every 15 min from min 60 through 120 during the clamp. Means were calculated using analysis of variance with fixed effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 120 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(GIR[0-120]) data.
Measure: Mean (Standard Deviation); unit: Grams per kilogram
Groups:
- Stage 2: Humulin Alone: Humulin-R: A single subcutaneous (SC) injection of 20 units (U)
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Grams per kilogram | 393 (242) | 597 (278) | 281 (123) | 637 (216)

12. Secondary Outcome: Area Under the Glucose Infusion Rate Curve From 0 to 180 Minutes After Injection (AUC[GIR{0-180}])
Description: The area under the curve for the glucose infusion rate from minutes (min) 0 to 180 after injection (AUC[GIR{0-180}]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) was measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 min prior to treatment, every 3 min from min 0 through 60, and every 15 min from min 60 through 180 during the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 180 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(GIR[180]) data.
Measure: Mean (Standard Deviation); unit: Grams per kilogram
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Grams per kilogram | 801 (420) | 1040 (501) | 604 (262) | 1150 (348)

13. Secondary Outcome: Area Under the Glucose Infusion Rate Curve From 0 to 240 Minutes After Injection (AUC[GIR{0-240}])
Description: The area the glucose infusion rate curve from minutes (min) 0 to 240 after injection (AUC[GIR{0-240}]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) was measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 min prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 to 240 during the clamp procedure. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose up to 240 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(GIR[240]) data.
Measure: Mean (Standard Deviation); unit: Grams per kilogram
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Grams per kilogram | 1240 (618) | 1430 (706) | 1010 (411) | 1630 (467)

14. Secondary Outcome: Area Under the Glucose Infusion Rate Curve From 0 to 360 Minutes After Injection (AUC[GIR{0-360}])
Description: The area under glucose infusion rate curve from minutes (min) 0 to 360 after injection (AUC[GIR{0-360}]) for participants who received Humalog or Humulin-R with or without recombinant human hyaluronidase (rHuPH20) was measured from blood samples obtained during a euglycemic clamp procedure. Samples were taken 10 and 1 min prior to treatment, every 3 min from min 0 through 60, every 15 min from min 60 through 180, and every 60 min from min 180 to 360 during the clamp. Means were calculated using analysis of variance with effects of participant, sequence within participant, treatment, and period.
Time Frame: Predose and up to 360 minutes postdose during Stage 1 or Stage 2
Population: Participants who received at least 1 dose of Humalog alone, Humalog + rHuPH20, Humulin-R alone, or Humulin-R + rHuPH20 with evaluable AUC(GIR[360]) data.
Measure: Mean (Standard Deviation); unit: Grams per kilogram
Groups:
- Stage 2: Humulin-R Alone: Humulin: A single subcutaneous (SC) injection of 20 units (U)
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Number analyzed (Participants) | 12 | 12 | 13 | 13
Grams per kilogram | 1940 (963) | 1930 (988) | 1860 (672) | 2260 (611)

ADVERSE EVENTS:
Description: AEs were classified by the body system affected.
Groups:
- Stage 1: Humalog Alone: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humalog alone during Stage 1 of the study
- Stage 1: Humalog + rHuPH20: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humalog + 300 U recombinant human hyaluronidase (rHuPH20) during Stage 1 of the study
- Stage 2: Humulin-R Alone: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humulin-R alone during Stage 2 of the study
- Stage 2: Humulin-R + rHuPH20: Participants randomized to treatment with a single subcutaneous (SC) injection of 20 units (U) Humulin-R + 240 U recombinant human hyaluronidase (rHuPH20) during Stage 2 of the study
Arm/Group | Stage 1: Humalog Alone | Stage 1: Humalog + rHuPH20 | Stage 2: Humulin-R Alone | Stage 2: Humulin-R + rHuPH20
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 2/13 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Humalog Alone (N=12) | Stage 1: Humalog + rHuPH20 (N=12) | Stage 2: Humulin-R Alone (N=13) | Stage 2: Humulin-R + rHuPH20 (N=14)
Infusion site pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza-like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.